CLINICAL TRIAL: NCT00895804
Title: Pharmacological Interaction Between Pindolol and MDMA (3,4-Methylenedioxymethamphetamine)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Heffter Research Institute (Other)
Responsible Party: Matthias E. Liechti, Universtity Hospital Basel
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: E-003/2001
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Mood Disorder; Substance-Related Disorders; Amphetamine-Related Disorders
Keywords: MDMA; beta adrenergic; Ecstasy
MeSH Terms: conditions — Mood Disorders; Substance-Related Disorders; Amphetamine-Related Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Pindolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pindolol, Placebo (Other): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two (actually 4) treatment conditions in the same subject.
  Interventions: Drug: MDMA; Drug: Pindolol
- MDMA, Placebo (Other): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two (actually 4) treatment conditions in the same subject.
  Interventions: Drug: MDMA; Drug: Pindolol

INTERVENTIONS:
Drug: MDMA — capsule, 1.6 mg/kg body weight, single dose
Drug: Pindolol — capsule of 20mg pindolol, single dose 1h before MDMA

SUMMARY:
MDMA (3,4-Methylenedioxymethamphetamine, "Ecstasy") produces tachycardia, hypertension, hyperthermia, and other acute adverse effects. Ecstasy use has also been associated with rare cardio- and cerebrovascular complications. The role of beta-blockers in the treatment of cardiovascular and adverse effects of MDMA is unknown.

DETAILED DESCRIPTION:
We investigated the interactive effects of the beta-blocker pindolol (20 mg) with MDMA (1.6 mg/kg) on heart rate, blood pressure, body temperature, and adverse effects in a double-blind placebo-controlled study in 16 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of the German language
* Subjects understand the procedures and the risks associated with the study
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids after midnight of the evening before the study session.
* Participants must be willing not to drive a traffic vehicle in the evening of the study day.
* Body mass index: 18-25 kg/m2

Exclusion Criteria:

* Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>140/90 mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder.
* Current or previous psychotic or affective disorder
* Psychotic or affective disorder in first-degree relatives
* Prior illicit drug use (except THC-containing products) more than 5 times or any time within the previous 2 months.
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2001-06; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Effect of pindolol on subjective response to MDMA | 24h

SECONDARY OUTCOMES:
Effect of pindolol on physiological response to MDMA | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Heffter Research Center, University Hospital of Psychiatry, Zurich, Canton of Zurich, Switzerland